CLINICAL TRIAL: NCT04515043
Title: AN EXPLORATORY FOLLOW-UP STUDY OF LONG TERM ANTI-TELOMERASE IMMUNE RESPONSE AFTER INVAC-1 VACCINATION IN PATIENTS WITH LONG TERM SURVIVAL. Addendum to INVAC1-CT-101 PROTOCOL - EUDRACT NUMBER : 2013-004369-15
Brief Title: EXPLORATORY STUDY Addendum to INVAC1-CT-101 (NCT02301754)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invectys (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INVAC1-CT-102
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INVAC-1 (Experimental): All patients have been treated by INVAC-1 vaccine during the previous phase 1 NCT02301754. No new treatment injection is required in this study.
  Interventions: Drug: INVAC-1 given in the previous phase 1 NCT02301754. No new injection is required in this study.

INTERVENTIONS:
Drug: INVAC-1 given in the previous phase 1 NCT02301754. No new injection is required in this study. — blood sampling will be drawn once in order to analyse long term memory immune response to INVAC-1 vaccine
  Other Names: blood sampling

SUMMARY:
This study will be an exploratory study of long term immunogenicity of INVAC-1 in patients who participated in the INVAC1-CT-101 phase I study (between 2014 and 2018).

DETAILED DESCRIPTION:
The primary goal of the study is to analyze anti-telomerase specific memory responses in blood of long term survival patients and to correlate these immune responses to their subsequent treatment since the end of INVAC1-CT-101 phase I study. Six patients are expected to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who participated in the phase I study and are still alive at the present time
2. Ability to provide written informed consent and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Anemia (Hgb < 7g/dL) according to L-1121-1 annexe 2 of Code de Santé Publique
2. Systolic blood pressure below 90 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
long term anti telomerase specific memory responses | 1 day visit
  will be measured by ELISPOT on blood of patients who were treated by INVAC-1 in the phase I NCT02301754 study and are still alive at the present time

CONTACTS AND LOCATIONS:
Overall Officials: Luis Teixeira, Principal Investigator — AP-HP Paris Hospital
Locations (1):
- Saint Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No